CLINICAL TRIAL: NCT01867099
Title: Long-term Outcome After Initially Successful Catheter Ablation of Atrial Fibrillation by Pulmonary Vein Isolation: a Ten-Year Cohort Study
Brief Title: Ten-year Outcomes After AF Ablation
Status: Completed | Type: Observational
Sponsor: Valley Health System (Other)
Responsible Party: Principal Investigator, Jonathan Steinberg,MD, Director, Arrhythmia Institute, Valley Health System
Other Study IDs: Valley 12.0032
Record Dates: First submitted 2013-05-29; First posted 2013-06-03 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Post-successful ablation: Patients who had undergone PVI ablation for AF and were free of AF for at least one year

SUMMARY:
Ablation of atrial fibrillation (AF) using pulmonary vein isolation is employed when patients do not respond favorably to medical therapy. Successful procedures are accomplished in the majority of patients, but the outcome after many years of follow-up after ablation is unknown.

DETAILED DESCRIPTION:
A prospectively identified cohort of 445 patients who demonstrated freedom from AF for at least one year following ablation (single procedure in 391, 87.9%) was followed for 66.0 ± 34.0 months. Patients were seen at least annually as outpatients, and underwent regular ECG monitoring, especially if there were symptoms suggestive of recurrent arrhythmia. Continued absence of arrhythmia was defined as freedom from AF or flutter > 30 secs.

ELIGIBILITY:
Inclusion Criteria:

* Prior AF ablation procedure
* No AF for one year post ablation

Exclusion Criteria:

* Geographic inaccessibility
* Longstanding persistent AF
* Recurrent AF within one year of ablation
* Prior AF ablation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent PVI ablation for drug refractory AF over a 10 year period and were free of AF for one year after last ablation procedure
Sampling Method: Non-Probability Sample
Enrollment: 445 (Actual)
Dates: Start 2002-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Atrial fibrillation or flutter > 30 secs | More than one year after successful primary ablation or redo procedure within 6 mos

CONTACTS AND LOCATIONS:
Locations (1):
- Valley Hospital, Ridgewood, New Jersey, United States